CLINICAL TRIAL: NCT05381090
Title: Circulating Ghrelin as a Biomarker for Dementia
Acronym: GDEM3
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Swansea University (Other)
Collaborators: Newcastle University (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Diagnostic
Other Study IDs: 288862
Record Dates: First submitted 2021-05-20; First posted 2022-05-19 (Actual); Last update posted 2023-10-26 (Actual); Status verified 2023-10

CONDITIONS: Dementia
MeSH Terms: conditions — Dementia

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (5):
- Healthy control (Active Comparator): Venous blood collection
  Interventions: Diagnostic Test: Venous blood collection
- Parkinson's disease (Experimental): Venous blood collection
  Interventions: Diagnostic Test: Venous blood collection
- Parkinson's disease dementia (Experimental): Venous blood collection
  Interventions: Diagnostic Test: Venous blood collection
- Dementia with Lewy Bodies (Experimental): Venous blood collection
  Interventions: Diagnostic Test: Venous blood collection
- Alzheimer's disease (Experimental): Venous blood collection
  Interventions: Diagnostic Test: Venous blood collection

INTERVENTIONS:
Diagnostic Test: Venous blood collection — Participants will undergo venous blood collection following an overnight fast and 5, 60 and 180 minutes following food intake.

SUMMARY:
The primary objective of this study will explore whether circulating acyl-ghrelin (AG) and unacylated-ghrelin (UAG) are reduced in neurodegenerative disease associated with cognitive impairment. It will focus on validating pilot data generated following the analysis of Parkinson's disease (PD), Parkinson's disease dementia (PDD) and healthy cohorts (IRAS project ID: 250933). In addition to the advantages of study replication we will extend the analysis to include two further patient groups that are associated with cognitive impairments, namely, Alzheimer's dementia (AD) and dementia with Lewy bodies (DLB). This study will increase confidence in the replication of our findings.

This will be a cross-sectional study using peripheral venous blood.

ELIGIBILITY:
Inclusion Criteria:

* Age > 60 years
* Subject or carer / legal representative is willing to sign consent document

Specific criteria for each group;

Parkinson's Disease

* PD diagnosed by a movement disorder specialist and meets the diagnosis of PD
* MoCA > 26/30
* No evidence of cognitive symptoms causing functional impairment

Parkinson's Disease Dementia

* PD diagnosed by a movement disorder specialist
* Duration of motor symptoms > 1 year
* Meets MDS task force criteria for PDD
* MoCA < 21/30

Dementia with Lewy Bodies

* Meets criteria for probable DLB as defined by the 4th report of the DLB consortium

Alzheimer's Disease

* Meets criteria for probable AD dementia (consistent with NIA/AA core clinical criteria for probable AD dementia)

Exclusion Criteria:

* Age < 60 years
* Current major depression
* Use of anti-psychotic medication
* Type I or Type II diabetes mellitus (DM) (excluding diet-controlled DM)
* Tobacco use
* BMI <15.0 kg/m2
* BMI > 30 kg/m2
* Comorbid gastrointestinal disease i.e. includes Coeliac, active Inflammatory Bowel Disease (Colitis), evidence for active gastric ulcers within the last 12 months, but excludes gastroesophageal reflux and hiatus hernia.
* >5 kg weight change over the preceding 3 months (determined by researcher from previous clinic visit and discussion with partner/carer)
* Significant active comorbidity
* Difficult venous access
* Vagotomy

Additional disease specific exclusions;

* Parkinson's Disease exclusion criteria
* Evidence of dementia or mild cognitive impairment
* Deep brain stimulation (DBS)
* Use of Duodopa

Parkinson's Disease Dementia exclusion criteria

* Dementia within 12 months of diagnosis of PD
* DBS

Dementia with Lewy bodies exclusion criteria

* Onset of motor Parkinsonism symptoms greater than 12 months prior to dementia diagnosis

Alzheimer's dementia exclusion criteria

* Presence of PD, PDD, DLB, or Frontotemporal Dementia (FTD)

Controls exclusion criteria

* Evidence of parkinsonism
* Evidence of dementia or mild cognitive impairment
* MoCA <26/30

Min Age: 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2022-08-15 (Actual); Primary Completion 2024-09 (Estimated); Study Completion 2024-09 (Estimated)

PRIMARY OUTCOMES:
Ghrelin ratio in PD and PDD | Through study completion, an average of 1 year
  Quantification of circulating ghrelin peptides

SECONDARY OUTCOMES:
Ghrelin ratio in AD and DLB | Through study completion, an average of 1 year
  Quantification of circulating ghrelin peptides

CONTACTS AND LOCATIONS:
Overall Officials: Jeffrey S Davies, BSc, PhD, Principal Investigator — Swansea University
Locations (1):
- Swansea University, Swansea, United Kingdom

IPD SHARING:
Plan to Share IPD: No